CLINICAL TRIAL: NCT05672810
Title: Correlation Between the Serum Level of Ferritin and D-dimer and the Severity of COVID-19 Infection
Brief Title: Serum Level of Ferritin and D-dimer and the Severity of (COVID 19) Infection
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Badawy AbdelFattah, Associate professor of chest diseases- Ain Shams University- Cairo- Egypt, Ain Shams University
Other Study IDs: FMASU MS220/2020
Record Dates: First submitted 2023-01-01; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: serum level of Ferritin and D-dimer — Blood venous sample

SUMMARY:
Many laboratory biomarkers were used for diagnosis of COVID-19 infection; however, their accuracy to assess the severity and prognosis are still to be evaluated.

Aim: to correlate between the serum Ferritin and D-dimer levels and the severity of COVID-19 infection and its outcome (mortality, days of hospital stay, ICU admission or mechanical ventilation).

A retrospective study conducted by retrieving patients' data who were admitted to Ain Shams University Specialized Hospital - Obour branch and diagnosed with COVID-19 infection in the period from 1st of April 2020 to 31st of July 2020.

DETAILED DESCRIPTION:
Aim of the study: to correlate between the serum level of Ferritin and D-dimer and the severity of COVID-19 infection as well as its outcome

Material and methods:

It is a retrospective study conducted by retrieving data of patients diagnosed with COVID-19 infection "PCR positive for SARS-CoV2" who were admitted to Ain Shams University Specialized Hospital - Obour branch in the period from 1st of April 2020 to 31st of July 2020.

The following data were collected from the studied patients' files:

• Demographic characteristics (age, sex, marital status, smoking status, co-morbidities), Source of infection, degree of severity of COVID-19 infection according to WHO Clinical management of COVID-19: interim guidance.

The investigations done include:

Laboratory investigations: including; (Complete blood picture, Iron profile, Liver function tests, D-dimer ("Using: using Biomerieux-VIDAS, Serial number IVD3002806, Manufactured in 2008, Marcy l'Étoile, France " "Reference range: 0-500 ng/ml") and Serum Ferritin ("using ABBOT-Architect 1000, Serial number I1SR62514, Manufactured in 2010, Chicago, Illinois, United States.""Reference range: 13-150 ng/ml" (Figure number "2") Radiological investigations: By High resolution CT chest ("Using: Toshiba 16-slice CT scanner, model number: activion 16, Manufactured in 2010, Japan") "severity scoring was done using "25-point CT severity score" Li et al, 2020". Score of 7 or less was considered as mild affection, 8-17 was considered as moderate affection and 18 or more was considered as severe affection " Saeed et al 2021"

Inclusion Criteria:

Hospitalized isolated patients "in Ain Shams University Specialized Hospital - Obour branch" with COVID-19 infection confirmed by "Polymerase chain reaction (PCR) positive for SARS-CoV2".

Exclusion Criteria:

* COVID-19 patients with other conditions altering the serum Ferritin level; For example; iron deficiency anemia, defective intestinal absorption, internal bleeding, rheumatoid arthritis, hyperthyroidism, leukemia, Hodgkin's lymphoma, frequent blood transfusions and advanced liver disease "Child-Pugh score C".
* COVID-19 patients with other conditions altering the serum D-dimer level; For example; known pulmonary embolism, known Deep Venous Thrombosis "DVT", pregnancy, heart failure, trauma, active malignancy, septicemia, disseminated Intra-vascular Coagulopathy "DIC".
* The patients with any missing studied data were also excluded. Data was correlated with the clinical spectrum of severity and the patient outcome regarding: death or recovery, days of hospital stay, need for ICU admission and need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized isolated patients "in Ain Shams University Specialized Hospital - Obour" with COVID-19 infection confirmed by "Polymerase chain reaction (PCR) positive for SARS-CoV2".

Exclusion Criteria:

* • COVID-19 patients with other conditions altering the serum Ferritin level; For example; iron deficiency anemia, defective intestinal absorption, internal bleeding, rheumatoid arthritis, hyperthyroidism, leukemia, Hodgkin's lymphoma, frequent blood transfusions and advanced liver disease "Child-Pugh score C".

  * COVID-19 patients with other conditions altering the serum D-dimer level; For example; known pulmonary embolism, known Deep Venous Thrombosis "DVT", pregnancy, heart failure, trauma, active malignancy, septicemia, disseminated Intra-vascular Coagulopathy "DIC".
  * The patients with any missing studied data were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is a retrospective study conducted by retrieving data of patients diagnosed with COVID-19 infection "PCR positive for SARS-CoV2" who were admitted to Ain Shams University Specialized Hospital - Obour
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Till study completion, an average of 4 months
Need for Mechanical ventilation | Till study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Eman B AbdelFattah, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication maybe shared
Supporting Information: Study Protocol, SAP
Time Frame: 3 months after publication
Access Criteria: Through the primary investigator e-mail to other interested researchers